CLINICAL TRIAL: NCT06103812
Title: Prospective, Multicentric, Observational Clinical Investigation to Evaluate the Performance and Safety of Hyalo4 Skin Gel in Management of Acute and Chronic Wounds.
Brief Title: Evaluate Performance and Safety of Hyalo4 Skin in Acute and Chronic Wounds
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Other Study IDs: AQG06-21-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Wound Heal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyalo4 Skin Gel
  Interventions: Device: Hyalo4 Skin Gel

INTERVENTIONS:
Device: Hyalo4 Skin Gel — The evaluation of performance and safety of Hyalo4 Skin Gel in the amelioration of bed wound appearance after 14 days of treatment.

SUMMARY:
Evaluate the performance and safety of the use of Hyalo4 Skin Gel in terms of wound management

DETAILED DESCRIPTION:
Ths clinical investigation study is to evaluate the performance and safety of Hyalo4 Skin Gel in the management of acute or chronic wounds of different etiology, according to the indication for use, the prescriptions of the clinicians and the standard procedures of the sites.

A maximum of 7 Visits will be performed, with the first 4 visits performed over a 4-weeks period for each patient and the last visit after 8 weeks from the first visit.

The schedule treatment will consist of daily medication changes, according to the instruction for use and the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Male or female ≥18 years.
3. Patients selected to be treated with Hyalo4 Skin Gel.
4. Patients with wound of the following etiology: first and second degree burns; surgical wounds; vascular ulcers; metabolic ulcers; pressure ulcers.
5. Patients followed on an outpatient or home basis.
6. Wound area ≥ 10 cm2 and ≤ 100 cm2

Exclusion Criteria:

1. Patients < 18 years.
2. Patients with acute or chronic infected lesions.
3. Hospitalized patients.
4. Women who are pregnant or breastfeeding or women who could become pregnant and are not using effective contraception.
5. Patients with acute or chronic lesions at high risk of infection, presenting at least one of the following criteria:

   * Stalled wound, without any clinical sign of healing progression
   * Immune system disorders
   * Protein-energy malnutrition
   * Alcohol, smoking and drug abuse (50ml of spirit, 0,5L of wine and 10 cigarettes/day)
   * Conditions associated with hypoxia and/or poor tissue perfusion
   * Corticosteroid, cytotoxic or immunosuppressive therapy.
6. Subjects unable to understand informed consent or having a high probability of non-compliance with the study procedures and or non-completion of the study according to investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or chronic wounds of different etiology (first and second degree burns; surgical wounds; vascular ulcers; metabolic ulcers; pressure ulcers),
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Performance of Hyalo4 Skin Gel treatment | 14 days
  The outcome will be measured as percentage of patients showing positive change in at least one of the following parameters: amelioration of wound tissue type (necrotic, slough, granulation tissue, epithelial tissue, closed), decrease of exudate amount (dry, moist, slightly exuding, heavily exuding, wet) and amelioration of exudate type (bloody, bloody/purulent, clear, murky, purulent, serous).

SECONDARY OUTCOMES:
EQ5D-Patient's quality of life | 56 days
  Patient's quality of life assessment will be evaluated as a change from baseline to 56 days after the start of treatment, through administration of EuroQoL-5D (EQ-5D).
Performance of treatment | 7,21,28,42 and 56 days
  The performance of Hyalo4 Skin Gel will be evaluated from baseline to 7, 21, 28, 42 and 56 days as amelioration of wound bed appearance in terms of: type of wound bed tissue and exudate quantity and quality.
Safety and Tollerability | 56 days
  The safety and tolerability of Hyalo4 Skin Gel will be assessed throughout all the visits by investigating local and expected adverse events, as consequence of the product application and any other adverse event occurred during the study.

CONTACTS AND LOCATIONS:
Locations (6):
- Slovakia (6):
  - Nemocnica Ružinov, Bratislava
  - BeneDerma s.r.o., Bratislava
  - Pedi-Derma s.r.o., Košice
  - POLIKLINIKA ProCare KVP, Košice
  - Nemocnica s poliklinikou Spišská Nová Ves, a.s., Spišská Nová Ves
  - Fakultná nemocnica s poliklinikou Žilina, Žilina

IPD SHARING:
Plan to Share IPD: Undecided